CLINICAL TRIAL: NCT05271071
Title: The Importance of Gluteus Maximus Muscle in Patients With Preliminary Diagnosis of Piriformis Syndrome: Prospective, Randomized, Single-Blind, Crossover Study
Brief Title: The Importance of Gluteus Maximus Muscle in Patients With Preliminary Diagnosis of Piriformis Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Bilge Cakir, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: IstanbulUC-BilgeCAKIR-1
Record Dates: First submitted 2022-02-18; First posted 2022-03-08 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Piriformis Muscle Syndrome; Myofacial Pain Syndromes; Piriformis Syndrome
Keywords: Piriformis Muscle Syndrome; Myofacial Pain Syndrome; Ultrasonography; Gluteus Maximus Muscle
MeSH Terms: conditions — Piriformis Muscle Syndrome; Facial Neuralgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gluteus Maximus Group (Active Comparator): 30 patients in the gluteus maximus group will be evaluated with detailed physical examination and special clinical tests. Sensitivity with sonopalpation, piriformis and gluteus maximus thicknesses, echo intensities will be evaluated with ultrasonography. Primarily diagnostic injection test for gluteus maximus muscle is planned for the first group with lidocaine with USG guide. At the first hour after injection full examination will be repeated for all patient and will be evaluated again with Numeric Rating Scale(NRS) at rest, with movement and with deep palpation. If the NRS score persists after the first injection patients will receive a diagnostic lidocaine injection into the piriformis muscle. At the first hour after the second injection, the physical examination and clinical tests of the patients will be repeated, and their pain at rest, with movement and with deep palpation will be evaluated with NRS.
  Interventions: Diagnostic Test: Ultrasound guided piriformis muscle and gluteus maximus muscle lidocaine injection
- Piriformis Muscle group (Active Comparator): 30 patients in the piriformis muscle group will be evaluated with detailed physical examination and special clinical tests. Sensitivity with sonopalpation, piriformis and gluteus maximus thicknesses, echo intensities will be evaluated with ultrasonography. Primarily diagnostic injection test for piriformis muscle (piriformis syndrome) is planned for the first group with lidocaine with USG guide. At the first hour after injection full examination will be repeated for all patient and will be evaluated again with Numeric Rating Scale(NRS) at rest, with movement and with deep palpation. If the NRS score persists after the first injection patients will receive a diagnostic lidocaine injection into the gluteus Maximus muscle. At the first hour after the second injection, the physical examination and clinical tests of the patients will be repeated, and their pain at rest, with movement and with deep palpation will be evaluated with NRS.
  Interventions: Diagnostic Test: Ultrasound guided piriformis muscle and gluteus maximus muscle lidocaine injection

INTERVENTIONS:
Diagnostic Test: Ultrasound guided piriformis muscle and gluteus maximus muscle lidocaine injection — Ultrasound guided piriformis muscle (piriformis syndrome) and gluteus maximus muscle 5 ml %1 lidocaine injection
  Other Names: Ultrasound guided piriformis muscle (piriformis syndrome) and gluteus maximus muscle (myofacial pain syndrome of gluteus Maximus muscle) diagnostic lidocaine injection

SUMMARY:
Literature shows different pathologies or combination pathologies can cause gluteal region pain and it can be difficult to diagnose. Piriformis syndrome is one of the cause of gluteal region pain, symptoms of myofascial pain syndrome affected gluteus maximus muscle may masquerade as piriformis muscle syndrome or both syndrome can be seen together. The aim of this study is diagnosis myofascial pain syndrome of gluteus maximus muscle and piriformis syndrome by physical examination, special clinical tests and ultrasound guided diagnostic injection test in patients presenting with gluteal pain and evaluate the coexistence of both syndromes.

DETAILED DESCRIPTION:
Piriformis syndrome is a painful clinical picture caused by entrapment of the sciatic nerve by the piriformis muscle at the exit of the pelvis, which causes pain in the gluteal region. It is characterized by symptoms of pain and numbness radiating from the thigh to the leg along the hip and sciatic trace. Compression/irritation of the sciatic nerve in or around the piriformis muscle constitutes the neuropathic component of the syndrome. Myofascial pain of the piriformis muscle is the primary cause of the somatic component of the syndrome. Various causes have been reported: congenital anomalies of piriformis muscle or sciatic nerve, trauma, overuse, muscle hypertrophy, shortening of the muscle, infection within the muscle, and leg length discrepancy. History, physical examination and ultrasound guided diagnostic injection test are key elements for the diagnosis.

Another cause of pain in the gluteal region is myofascial pain syndrome of gluteus maximus muscle. Myofascial pain syndrome is a largely underdiagnosed and undertreated entity. Prevalence varies from 30 to 93% among the persons with musculoskeletal pain. Myofascial pain syndrome is a syndrome characterized by acute or chronic regional pain originating from localized trigger points in the muscle and fascia. Traumatic events, muscular overloads, psychological stress, and systemic pathology may lead to development of one or more palpable bands or trigger points. Myofascial pain syndrome affecting the gluteus maximus muscle causes pain in the medial and lower parts of the muscle; It is characterized by pain that usually radiates throughout the hip and sometimes into the coccygeal region. The diagnosis of myofascial pain syndrome is based on a pertinent history and physical examination.

The purpose of the study is; to evaluate the myofascial pain syndrome of gluteus maximus muscle and piriformis syndrome with physical examination, special clinical tests, ultrasonographic examinations and, to confirm the presence of myofascial pain syndrome of gluteus maximus muscle accompanying piriformis syndrome with the evaluation of clinical findings after the gluteus maximus and piriformis muscle diagnostic injections.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* Had unilateral hip pain and/or leg pain
* Had Positive trigger point or taut band or pain with pression in piriformis muscle
* Patients whose informed consent was obtained for participation in the study

Exclusion Criteria:

* History of hip surgery
* History of spinal surgery
* Clinical diagnosis of Inflammatory rheumatic diseases
* History of spinal or pelvic fracture
* Clinical diagnosis of osteoarthritis or history of fracture of the lower extremities
* Had uncontrolled diabetes
* Pregnancy or breastfeeding
* Had allergy to lidocaine
* Had gluteal injection in the previous 6 months
* Had anticoagulant or antiplatelet treatment
* Had skin infection at the site of needle entry
* Had radiculopathy caused by lumbar disc pathology
* Had neurological disease
* Tumors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Pain via Numeric Rating Scale at 60 Minutes after piriformis muscle/gluteus maximus Injection (first injection) | Baseline, 60 minutes after gluteus maximus injection, 60 minutes after piriformis muscle injection.
  Pain of the participants will be assessed by one of the most commonly used pain scale "numerical rating scale". It is numeric version of visual analog scale in which a patient selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing "no pain" to '10' representing "pain as bad as you can imagine". Participant is asked to indicate rates of their pain on the day of presentation during resting, during function and physical examination as a baseline and, 60 minutes after gluteus maximus injection for each, 60 minutes after piriformis muscle injection for each.

SECONDARY OUTCOMES:
Change from Baseline Pain via Numeric Rating Scale at 60 Minutes after Second Injection | Baseline, 60 minutes after gluteus maximus injection, 60 minutes after piriformis muscle injection.
  Pain of the participants will be assessed by one of the most commonly used pain scale "numerical rating scale". It is numeric version of visual analog scale in which a patient selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing "no pain" to '10' representing "pain as bad as you can imagine". Participant is asked to indicate rates of their pain on the day of presentation during resting, during function and physical examination as a baseline and, 60 minutes after gluteus maximus injection for each, 60 minutes after piriformis muscle injection for each.

CONTACTS AND LOCATIONS:
Overall Officials: Bilge Cakir, Principal Investigator — Istanbul University - Cerrahpasa; Kenan Akgun, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University- Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Probst D, Stout A, Hunt D. Piriformis Syndrome: A Narrative Review of the Anatomy, Diagnosis, and Treatment. PM R. 2019 Aug;11 Suppl 1:S54-S63. doi: 10.1002/pmrj.12189. Epub 2019 Jul 22. PMID 31102324
- [Background] Kirschner JS, Foye PM, Cole JL. Piriformis syndrome, diagnosis and treatment. Muscle Nerve. 2009 Jul;40(1):10-8. doi: 10.1002/mus.21318. PMID 19466717
- [Background] Cass SP. Piriformis syndrome: a cause of nondiscogenic sciatica. Curr Sports Med Rep. 2015 Jan;14(1):41-4. doi: 10.1249/JSR.0000000000000110. PMID 25574881
- [Background] Hopayian K, Danielyan A. Four symptoms define the piriformis syndrome: an updated systematic review of its clinical features. Eur J Orthop Surg Traumatol. 2018 Feb;28(2):155-164. doi: 10.1007/s00590-017-2031-8. Epub 2017 Aug 23. PMID 28836092
- [Background] Hopayian K, Song F, Riera R, Sambandan S. The clinical features of the piriformis syndrome: a systematic review. Eur Spine J. 2010 Dec;19(12):2095-109. doi: 10.1007/s00586-010-1504-9. Epub 2010 Jul 3. PMID 20596735
- [Background] Jankovic D, Peng P, van Zundert A. Brief review: piriformis syndrome: etiology, diagnosis, and management. Can J Anaesth. 2013 Oct;60(10):1003-12. doi: 10.1007/s12630-013-0009-5. Epub 2013 Jul 27. PMID 23893704
- [Background] Hermann W. [The piriformis syndrome-a special indication for botulinum toxin]. Nervenarzt. 2020 Feb;91(2):99-106. doi: 10.1007/s00115-020-00866-4. German. PMID 32020236
- [Background] Kuncewicz E, Gajewska E, Sobieska M, Samborski W. Piriformis muscle syndrome. Ann Acad Med Stetin. 2006;52(3):99-101; discussion 101. PMID 17385355
- [Background] Siddiq MA, Hossain MS, Uddin MM, Jahan I, Khasru MR, Haider NM, Rasker JJ. Piriformis syndrome: a case series of 31 Bangladeshi people with literature review. Eur J Orthop Surg Traumatol. 2017 Feb;27(2):193-203. doi: 10.1007/s00590-016-1853-0. Epub 2016 Sep 19. PMID 27644428
- [Background] Borg-Stein J, Iaccarino MA. Myofascial pain syndrome treatments. Phys Med Rehabil Clin N Am. 2014 May;25(2):357-74. doi: 10.1016/j.pmr.2014.01.012. Epub 2014 Mar 17. PMID 24787338
- [Background] Money S. Pathophysiology of Trigger Points in Myofascial Pain Syndrome. J Pain Palliat Care Pharmacother. 2017 Jun;31(2):158-159. doi: 10.1080/15360288.2017.1298688. Epub 2017 Apr 5. PMID 28379050
- [Background] Saxena A, Chansoria M, Tomar G, Kumar A. Myofascial pain syndrome: an overview. J Pain Palliat Care Pharmacother. 2015 Mar;29(1):16-21. doi: 10.3109/15360288.2014.997853. Epub 2015 Jan 5. PMID 25558924
- [Background] Gerwin RD. Diagnosis of myofascial pain syndrome. Phys Med Rehabil Clin N Am. 2014 May;25(2):341-55. doi: 10.1016/j.pmr.2014.01.011. Epub 2014 Mar 18. PMID 24787337